CLINICAL TRIAL: NCT01446367
Title: Corneal Topographic Changes After 20-gauge Pars Plana Vitrectomy Associated With Scleral Buckling for the Treatment of Rhegmatogenous Retinal Detachment
Brief Title: Corneal Changes After Retinal Surgery
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Alexandre Grandinetti, Principal Investigator, Universidade Federal do Paraná
Other Study IDs: Cornea vs Vit-buckle
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Rhegmatogenous Retinal Detachment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the corneal changes after performing 20 gauge vitrectomy associated with scleral buckling for the treatment of rhegmatogenous retinal detachment.

DETAILED DESCRIPTION:
Patients submitted to 20-gauge vitrectomy associated with scleral buckling were evaluated with corneal topography before surgery and in the 7,30 and 90 days after surgery to asses corneal curvature changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rhegmatogenous retinal detachments

Exclusion Criteria:

* Previous eye surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rhegmatogenous retinal detachments
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

REFERENCES:
- [Background] Weinberger D, Lichter H, Loya N, Axer-Siegel R, Muzmacher L, Gabbay U, Yassur Y. Corneal topographic changes after retinal and vitreous surgery. Ophthalmology. 1999 Aug;106(8):1521-4. doi: 10.1016/S0161-6420(99)90447-5. PMID 10442898